CLINICAL TRIAL: NCT04305041
Title: A Phase 1/2 Open-label Rolling-arm Umbrella Platform Design of Investigational Agents With or Without Pembrolizumab or Pembrolizumab Alone in Participants With Melanoma (KEYMAKER-U02): Substudy 02A
Brief Title: Substudy 02A: Safety and Efficacy of Pembrolizumab in Combination With Investigational Agents in Participants With Programmed Cell-death 1 (PD-1) Refractory Melanoma (MK-3475-02A/KEYMAKER-U02)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-02A; MK-3475-02A (Other: MSD); KEYMAKER-U02 (Other: MSD); 2023-506312-41-00 (Registry Identifier: EU CT); U1111-1293-5630 (Registry Identifier: UTN); 2019-003956-35 (EudraCT Number)
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
Keywords: receptor tyrosine kinase inhibitor; programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); T cell immunoreceptor with immunoglobulin and immunoreceptor tyrosine receptor motif domains (TIGIT)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab + Quavonlimab + Vibostolimab (Experimental): Participants will receive pembrolizumab intravenously (IV) plus quavonlimab IV plus vibostolimab IV at specified doses on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Pembrolizumab; Biological: Quavonlimab; Biological: Vibostolimab
- Pembrolizumab + Quavonlimab + Lenvatinib (Experimental): Participants will receive pembrolizumab IV plus quavonlimab IV plus lenvatinib orally at specified doses on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Pembrolizumab; Biological: Quavonlimab; Drug: Lenvatinib
- Pembrolizumab + all-trans retinoic acid (ATRA) (Experimental): Participants will receive pembrolizumab IV plus ATRA orally at specified doses on specified days for a total treatment duration of up to approximately 2 years
  Interventions: Drug: ATRA

INTERVENTIONS:
Biological: Pembrolizumab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + Quavonlimab + Lenvatinib; Pembrolizumab + Quavonlimab + Vibostolimab
Biological: Quavonlimab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-1308
  Arms: Pembrolizumab + Quavonlimab + Lenvatinib; Pembrolizumab + Quavonlimab + Vibostolimab
Biological: Vibostolimab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-7684
  Arms: Pembrolizumab + Quavonlimab + Vibostolimab
Drug: Lenvatinib — Administered via oral capsules at a specified dose on specified days
  Other Names: MK-7902; LENVIMA®
  Arms: Pembrolizumab + Quavonlimab + Lenvatinib
Drug: ATRA — Administered via oral capsules at a specified dose on specified days
  Other Names: VESANOID
  Arms: Pembrolizumab + all-trans retinoic acid (ATRA)

SUMMARY:
Substudy 02A is part of a larger research study that is testing experimental treatments for melanoma, a type of skin cancer. The larger study is the umbrella study.

The goal of substudy 02A is to evaluate the safety and efficacy of investigational treatment arms in participants with PD-1 refractory melanoma to identify the investigational agent(s) that, when used in combination, are superior to the current treatment options/historical control available.

As of Amendment 4 (effective date: 05JAN2022), a third arm has been opened to participant enrollment, treatment with pembrolizumab and all-trans retinoic acid (ATRA). Enrollment into the first two arms, treatment with pembrolizumab + quavonlimab+ vibostolimab and treatment with pembrolizumab + quavonlimab + lenvatinib has been completed per protocol as of September 2021.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed melanoma
* Has unresectable Stage III or Stage IV melanoma, not amenable to local therapy
* Has progressed on treatment with an anti-PD-1/L1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other therapies
* Has imaging documenting progression per RECIST 1.1 and iRECIST after initiation of an anti-PD-1/L1 agent, or by RECIST 1.1 if progression occurred on adjuvant therapy or in the setting of rapid progression.
* Has not received more than 3 lines of therapy for their advanced melanoma
* Has provided a tumor biopsy
* Male participants who receive lenvatinib or ATRA are abstinent from heterosexual intercourse or agree to use contraception during the intervention period and for at least 7 days after the last dose of lenvatinib or ATRA; for male participants who only receive pembrolizumab, quavonlimab, vibostolimab, or a combination, no contraception measures are needed
* Female participant are not pregnant or breastfeeding and are either not a woman of child-bearing potential (WOCBP) OR use a contraceptive method that is highly effective or are abstinent from heterosexual intercourse during the intervention period and for at least 120 days after the last dose of pembrolizumab, quavonlimab, vibostolimab or 30 days after the last dose of lenvatinib or ATRA, whichever occurs last
* Has adequate organ function
* Has resolution of toxic effect(s) of the most recent prior therapy to Grade 1 or less (except alopecia)

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving immunosuppressive therapy within 7 days before the first dose of study intervention
* Has a known additional malignancy that is progressing or requires active treatment within the past 2 years
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has ocular or mucosal melanoma
* Has known hypersensitivity including previous clinically significant hypersensitivity reaction to treatment with another mAb
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has an active infection requiring systemic therapy
* Has known history of human immunodeficiency virus (HIV)
* Has known history of hepatitis B
* Has a history of (noninfectious) pneumonitis
* Has a history of active tuberculosis (TB)
* Has received prior systemic anticancer therapy within 4 weeks prior to randomization
* Has received prior radiotherapy within 2 weeks of first dose of study intervention
* Has had major surgery <3 weeks prior to first dose of study intervention
* Has received a live vaccine within 30 days before the first dose of study intervention
* Has participated in a study of an investigational agent within 4 weeks prior to the first dose of study intervention
* Has had an allogeneic tissue/solid organ transplant
* Has a pre-existing Grade ≥3 gastrointestinal fistula or nongastrointestinal fistula
* Has radiographic evidence of encasement of invasion of major blood vessel or of intratumoral cavitation
* Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study intervention
* Has clinically significant cardiovascular disease within 12 months from first dose of study intervention

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who experience an adverse event (AE) | Up to ~28 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience an AE will be reported.
Percentage of participants who discontinue study treatment due to an AE | Up to ~24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinue study treatment due to an AE will be reported.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) | Up to ~30 months
  ORR is defined as the percentage of participants in the analysis population who have a complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters). Responses are according to RECIST 1.1 as assessed by blinded independent central review (BICR). RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ.

SECONDARY OUTCOMES:
Duration of Response (DOR) per RECIST 1.1 | Up to ~30 months
  For participants in the analysis population who show a confirmed CR (disappearance of all target lesions) or confirmed PR (at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters), DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death due to any cause, whichever occurs first. Responses are according to RECIST 1.1 as assessed by BICR. RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (36):
- United States (13):
  - The Angeles Clinic and Research Institute ( Site 1009), Los Angeles, California
  - UCLA Hematology & Oncology ( Site 1004), Los Angeles, California
  - Providence Saint John's Health Center ( Site 1010), Santa Monica, California
  - University of Colorado, Anschutz Cancer Pavilion ( Site 1012), Aurora, Colorado
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins ( Site 1022), Baltimore, Maryland
  - NYU Clinical Cancer Center ( Site 1002), New York, New York
  - Duke Cancer Institute ( Site 1005), Durham, North Carolina
  - Martha Morehouse Tower ( Site 1020), Columbus, Ohio
  - Oregon Health & Science University ( Site 1013), Portland, Oregon
  - University of Pennsylvania Abramson Cancer Center ( Site 1008), Philadelphia, Pennsylvania
  - West Cancer Center - East Campus ( Site 1014), Germantown, Tennessee
  - University of Texas MD Anderson Cancer Center ( Site 1006), Houston, Texas
  - Inova Schar Cancer Institute ( Site 1011), Fairfax, Virginia
- Australia (4):
  - Calvary Mater Newcastle-Medical Oncology ( Site 1404), Waratah, New South Wales
  - Melanoma Institute Australia ( Site 1402), Wollstonecraft, New South Wales
  - Tasman Oncology Research Pty Ltd ( Site 1403), Southport, Queensland
  - Fiona Stanley Hospital ( Site 1401), Murdoch, Western Australia
- France (6):
  - Hopital La Timone ( Site 1103), Marseille, Bouches-du-Rhone
  - Hopital Saint Andre ( Site 1108), Bordeaux, Gironde
  - Institut Claudius Regaud ( Site 1105), Toulouse, Haute-Garonne
  - Centre Hospitalier Lyon Sud ( Site 1102), Pierre-Bénite, Rhone
  - A.P.H. Paris, Hopital Saint Louis ( Site 1107), Paris
  - Gustave Roussy ( Site 1101), Villejuif, Île-de-France Region
- Israel (4):
  - HaEmek Medical Center ( Site 1703), Afula
  - Rambam Health Care Campus-Oncology ( Site 1704), Haifa
  - Hadassah Ein Karem Jerusalem ( Site 1702), Jerusalem
  - Chaim Sheba Medical Center ( Site 1701), Ramat Gan
- Italy (5):
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 1399), Milan
  - Istituto Europeo di Oncologia ( Site 1301), Milan
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 1302), Napoli
  - Istituto Oncologico Veneto IRCCS ( Site 1355), Padua
  - Policlinico Le Scotte - A.O. Senese ( Site 1377), Siena
- CANCERCARE LANGENHOVEN DRIVE ONCOLOGY CENTRE-Clinical Trials Unit ( Site 1865), Port Elizabeth, Eastern Cape, South Africa
- Switzerland (3):
  - Hôpitaux Universitaires de Genève (HUG)-Oncology ( Site 1603), Geneva, Canton of Geneva
  - CHUV Centre Hospitalier Universitaire Vaudois ( Site 1602), Lausanne, Canton of Vaud
  - Universitaetsspital Zuerich ( Site 1601), Zuerich Flughafen, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26249&tenant=MT_MSD_9011